CLINICAL TRIAL: NCT04132596
Title: Non-invasive Spinal Cord Stimulation Combined With Activity-based Rehabilitation in Chronic Spinal Cord Injury
Brief Title: Spinal Stimulation in Chronic Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Neurokinex Charitable Trust (Other)
Collaborators: International Spinal Research Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pathfinder 2.0
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Motor Complete Tetraplegia (Experimental): C4-T1 American Spinal Injuries Association (ASIA) Impairment Scale Classification A or B spinal cord injury tscs with activity based therapy intervention
  Interventions: Device: Transcutaneous spinal cord stimulation; Other: Activity Based Therapy
- Motor Complete Paraplegia (Experimental): T2-12 ASIA Impairment Scale A or B spinal cord injury tscs with activity based therapy intervention
  Interventions: Device: Transcutaneous spinal cord stimulation; Other: Activity Based Therapy
- Motor incomplete SCI (Experimental): C4-T12 ASIA Impairment Scale C or D spinal cord injury tscs with activity based therapy intervention
  Interventions: Device: Transcutaneous spinal cord stimulation; Other: Activity Based Therapy

INTERVENTIONS:
Device: Transcutaneous spinal cord stimulation — Electrical stimulation of the spinal cord via transcutaneous hydrogel electrodes
Other: Activity Based Therapy — Physical therapy

SUMMARY:
Electrical spinal stimulation combined with activity-based rehabilitation (ABR) can improve motor and autonomic function in individuals suffering from varying degrees of paralysis. Spinal stimulation studies have included invasive implanted devices and non-invasive transcutaneous systems using different combinations of stimulation current, waveform, amplitude, duration and spinal levels targeted. Invasive and non-invasive systems have been demonstrated to permit individuals with chronic spinal cord injury (SCI), previously considered to have complete injuries on the International Standards for the Neurological Classification of Spinal Cord Injuries (ISNCSCI) scale (Classification A), to regain some degree of voluntary and autonomic function during periods of stimulation. The aim of this study is to evaluate the effects of a novel non-invasive transcutaneous electrical spinal cord stimulation system (tSCS) combined with activity-based rehabilitation in patients who have paralysis of their legs and/or arms. We will examine participants for any changes in sensory, motor or autonomic function. We will use a transcutaneous spinal cord stimulator that has been designed to deliver safe and tolerable bursts of high frequency pulsed current that minimise the capacitance efforts of the skin surface and maximise conductance of a second waveform using low frequency current to target neural structures. We aim to investigate this form of neuromodulation with a small group of individuals with chronic spinal cord injury. Our goal is to observe and describe any short term or lasting changes in function that can safely and comfortably be derived from this combination of spinal stimulation and activity-based rehabilitation. If this therapy can cause lasting improvements in sensory, motor, respiratory or autonomic function, then this may lead to a greater degree of functional independence for these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Aged 18 years or over
* Injury level C4-T12
* At least one year post spinal cord injury
* Medically stable and cognitively intact
* Independent respiration, not requiring any ventilatory support

Exclusion Criteria:

* Any active implanted metallic device including, but not limited to neurostimulators, cochlear implants, pacemakers, implantable defibrillators or drug delivery pump
* Implanted surgical hardware that is not compatible with MRI scanners
* Possible, suspected or confirmed pregnancy and/or lactation
* Active Heterotopic Ossification
* Recent history or fracture, contractures or pressure sore, deep vein thrombosis or urinary tract or other infection that may interfere with the intervention and training.
* History of epilepsy and/or seizures.
* Severe spasticity which have been unstable over the past 3 months prior to enrolment and not expected to change; taking varying doses of anti-spasticity medications which could not be tapered to a stable dose and is not expected to change
* Botulinum toxin injections within 6 months of participation (excluding bladder)
* Non-injury related neurological impairment
* Clinically significant severe depression in spite of treatment
* Patients who have cardiovascular disease
* Patients with Autonomic Dysreflexia that is severe, ongoing and has required medical treatment within the past one month
* Active aggressive tumour within or surrounding the spinal cord or brain stem
* A syrinx (fluid filled cavity) in the spinal cord
* Skin conditions or allergies that may affect electrode placement
* Bodyweight over 120kg (due to inability to use some of the study equipment)
* Patients who do not understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
International Standards for the Neurological Classification of Spinal Cord Injury Classification scores (ISNCSCI ASIA chart) | 1 year
  Sensory and motor scores. Sensory scale 0-224, motor scale 0-100 with higher scores relating to increased sensation and motor power
Spinal Cord Independence Measure (SCIM) | 1 year
  Functional independence tool for spinal cord injury. Scale of 0-100, with higher scores meaning increased function
Berg Balance Score (where applicable) | 1 year
  Measure of standing balance. Scale of 0-56, with higher values meaning increased standing balance and reduced risk of falls
NeuroRecovery Scale (NRS) | 1 year
  Functional independence measure rated from 1a, the lowest classification of functioning to 4C, the highest classification of functioning
Graded Redefined Assessment of Strength, Sensation and Prehension (GRASSP) Test | 1 year
  Upper limb measure of sensation and function. Strength scored 0-100, sensation scored 0-24 and prehension scored 0-64. Increased score relates to increased hand strength, sensation and function
Capabilities of Upper Extremity Questionnaire (CUE) | 1 year
  Upper limb capability questionnaire with 32 items. Scores between 32-124 with higher scores associated with higher levels of function of the upper limb
Force dynamometry - hand | 1 year
  Grip and pinch strength using JTech force transducers. Measurements taken in Newtons
Electromyography (EMG) of muscle activity | 1 year
  Upper limb, trunk and lower limb EMG using the Delsys Trigno System

SECONDARY OUTCOMES:
World Health Organisation Quality Of Life - BREF (WHOQOL-BREF) | 1 year
  Quality of Life self report questionnaire with 26 items, subdivided into Physical Health (raw score range 7-35), Psychological Health (raw score range 6-30), Social Relationships (raw score range 3-15), Environment (raw score range 8-40)
International Spinal Cord Society Autonomic Standards Assessment Form | 1 year
  Bladder function questionnaire to document method of bladder management
International Spinal Cord Society Autonomic Standards Assessment Form | 1 year
  Bowel function questionnaire to document method of bowel management
International Spinal Cord Society Autonomic Standards Assessment Form | 1 year
  Cardiovascular function questionnaire to document ability to regulate cardiovascular system
International Spinal Cord Society Autonomic Standards Assessment Form | 1 year
  Sexual function questionnaire to document symptoms and impairments resulting from spinal cord injury
Modified Ashworth Scale | 1 year
  Spasticity measure, scores of 0 - no increase in spasticity to 4 - affected part rigid
Respiratory function tests of maximal inspiratory and expiratory pressures | 1 year
  Maximal inspiratory and expiratory pressures in breathing,

CONTACTS AND LOCATIONS:
Overall Officials: Jane Symonds, Physio, Principal Investigator — Clinical Lead Physiotherapist
Locations (2):
- United Kingdom (2):
  - Neurokinex, Gatwick
  - Neurokinex, Hemel Hempstead

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suggitt J, Symonds J, D'Amico JM. Safety and Effectiveness of Multisite Transcutaneous Spinal Cord Stimulation Combined With Activity-Based Therapy When Delivered in a Community Rehabilitation Setting: A Real-World Pilot Study. Neuromodulation. 2025 Oct;28(7):1144-1156. doi: 10.1016/j.neurom.2025.01.005. Epub 2025 Feb 24. PMID 39998450
- See also: Related Info — http://www.neurokinex.org